CLINICAL TRIAL: NCT04723407
Title: Assessment of the Psychological Impact of the COVID19 (SARS-CoV-2) Pandemic on Patients With Chronic Inflammatory Rheumatism According to a Management Strategy in the Rheumatology Department of Limoges University Hospital
Brief Title: Assessment of the Psychological Impact of the COVID19 (SARS-CoV-2) Pandemic on Patients With Chronic Inflammatory Rheumatism
Acronym: RICOVID19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI20_0062 /RICOVID19
Record Dates: First submitted 2021-01-22; First posted 2021-01-25 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Rheumatism
MeSH Terms: conditions — Rheumatic Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed patients: Those who had the management strategy implemented by the service during confinement
  Interventions: Other: questionnaires
- Unexposed patients: Those who could not benefit from this strategy
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Questionnaire completion

SUMMARY:
Patients with chronic inflammatory rheumatism (RIC) or autoimmune diseases, rheumatoid arthritis and spondyloarthritis, are regularly monitored in consultation as part of a "treat to target" strategy with rapid adaptation of treatments to the activity of their disease. according to French recommendations.

They are treated with immunosuppressive drugs: disease-modifying treatments with very often methotrexate, associated with biotherapies or targeted therapies (JAK inhibitors) They can also be treated transiently or over the long term with corticosteroids. These treatments expose them to greater infectious risks, especially with regard to COVID19.

The objective is on the one hand to assess the impact of the Covid 19 pandemic on general state of health of these patients and the evolution of their disease and on the other hand to prioritize the optimal care of these patients by including in the context of maintaining the pandemic reduction rules, modern telemedicine technologies.

ELIGIBILITY:
Inclusion Criteria:

All patients with chronic inflammatory rheumatism followed in the rheumatology department of the CHU de Limoges.

Exclusion Criteria:

Patients who object to the use of their data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic inflammatory rheumatism followed in the rheumatology department of the CHU de Limoges
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
post-traumatic stress | Day 1
  Presence or absence of post-traumatic stress disorder due to the COVID19 pandemic assessed by the Post-traumatic stress disorder Check-list version DSM-5 (PCL-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Département de Rhumatologie, Limoges, France